CLINICAL TRIAL: NCT00058903
Title: Treatment of Cholestatic Pruritus With Sertraline
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRCPWS (completed)
Record Dates: First submitted 2003-04-14; First posted 2003-04-16 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Pruritus; Liver Cirrhosis, Biliary; Hepatitis C
Keywords: Cholestatic; Pruritus; Sertraline; primary biliary cirrhosis; hepatitis C
MeSH Terms: conditions — Pruritus; Liver Cirrhosis, Biliary; Hepatitis C | interventions — Sertraline

INTERVENTIONS:
Drug: sertraline

SUMMARY:
The goal of this study is to find an effective and well-tolerated medical therapy for itching due to liver disease. Persons with primary biliary cirrhosis or chronic hepatitis C are currently being enrolled in the study. Persons participating in the study are given sertraline, a medication which is also often used for depression,to treat their itching. The dose is gradually increased as the effect on itching and any other potential side effects are carefully monitored.

ELIGIBILITY:
* Itching for at least 3 months
* Primary biliary cirrhosis or hepatitis C
* Elevated alkaline phosphatase for at least 6 months

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2003-04; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States